CLINICAL TRIAL: NCT04895683
Title: Can Behavioural-science Informed Text Messages Improve COVID-19 Vaccination Uptake in North West London? A RCT
Brief Title: Using Text Messages to Improve COVID-19 Vaccination Uptake
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Central London CCG (Unknown); Imperial College Health Partners (Unknown); Institute for Global Health Innovations (Unknown); The Behavioural Insights Team (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21SM6815
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: text message; vaccination; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: 3-armed parallel randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: The researcher conducting the data analysis will do so using a trial arm code. They will not have the key to unlock which trial arm is which.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - Control SMS (Active Comparator): Control (current practice) text message invitation
  Interventions: Behavioral: Text message content
- Arm 2 - Behavioural Science informed SMS content (Experimental): Experimental text message invitation
  Interventions: Behavioral: Text message content
- Arm 3 - Pre-alert and behavioural science informed SMS content (Experimental): Two text messages, including a pre-alert SMS and the text message intervention in trial arm 2.
  Interventions: Behavioral: Text message content

INTERVENTIONS:
Behavioral: Text message content — Behavioural science-informed text messages aimed at improving COVID-19 vaccination uptake.

SUMMARY:
COVID-19 vaccinations significantly reduce the risk of getting seriously ill or dying from COVID-19. Since December 2020, the UK has rolled out vaccinations according to the Joint Committee for Vaccinations and Immunity (JCVI) priority groups. However, despite data indicating that more than 90% of the UK population intends to get vaccinated, there are geographical and ethnic variations in vaccination acceptance. As younger cohorts with lower risk from COVID-19 become eligible for vaccination, it is expected that uptake rates may also be lower than they have been in previous cohorts.

It was recently announced that a national NHS text message service will be introduced to invite individuals eligible for the COVID-19 vaccine to book a vaccination appointment. Many GP practices and CCGs have already implemented text messages to invite eligible residents and patients for the vaccine.

However, recent research has shown that the message content of text messages inviting members of the public to other preventative health opportunities (e.g. personalised messages and GP-endorsements in cancer screening) can impact uptake.

This 3-arm randomised controlled trial will be conducted across the Central London (CL) Clinical Commissioning Group (CCG) which to-date has seen the lowest rates of COVID-19 vaccination uptake in the country. The study aims to investigate the most effective text message strategy to inform local, regional and national practice.

The intervention text message content to be tested is informed by behavioural science theory is personalised to include the recipient's name and GP practice name. All patients in the Central London CCG who are unvaccinated, aged 18-49, who have not declined the vaccine will be included as their cohort becomes eligible for vaccination according to the JCVI guidelines. The trial will compare the uptake of the COVID-19 vaccination by trial arm at 3 and 8 weeks after the intervention is deployed.

DETAILED DESCRIPTION:
The COVID-19 vaccine is an effective way to reduce morbidity and mortality from COVID-19. Increasing uptake of the COVID-19 vaccine is a major public health priority. People's willingness to receive the COVID- 19 vaccine in the UK has been at record highs - 9 in 10 people said they would receive it when the NHS notifies them that it is their turn. However, evidence suggests that willingness to get vaccinated is lower amongst younger age groups and BAME populations. Additionally, high willingness to be vaccinated may not translate into high uptake, particularly as the vaccine rollout extends to younger, less vulnerable cohorts.

Uptake of the COVID-19 vaccine may be influenced by many factors, including personal beliefs such as perceived low personal risk from COVID-19, perceived social and cultural norms or a concerns around vaccine safety or efficacy. Additionally, process barriers, such as the effort required to attend an appointment may reduce vaccine uptake. With more than 95% of UK households having a mobile phone, text messages can be an effective way to improve uptake of healthcare services and medicine adherence. In particular, recent research has shown that reminder text messages about flu vaccination appointments can improve uptake by up to 10%, and that some messages may be more effective for specific groups. However, more research is needed to maximise the effectiveness of messages to increase uptake of the COVID-19 vaccine specifically and to explore how the effectiveness of messaging differs across different age and ethnicity groups.

The proposed research will determine which message strategy increases COVID-19 vaccine vaccination rates in the cohort aged between 18 and 49 years old as they become eligible for the vaccine according to JCVI categories.

During the trial, each cohort that newly becomes eligible to be vaccinated will be randomised to one of the five trial text message strategies.

The trial arms will include the current practice text message invitation which will act as the control and four intervention trial arms. The intervention text message strategies and message content have been based on behavioural science theory.

The usual care team will deploy the text messages according to the trial arm allocation. The vaccination status will be recorded in the patients electronic health record (EHR) as per usual practice. Researchers will have access to the pseudonymised datasets through a secure data platform which only holds pseudonomised data (see data Study Procedure section).

Analysis will measure and compare the vaccination uptake across trial arms.

ELIGIBILITY:
Inclusion Criteria:

* Residents registered with a GP practice in the Central London (Westminster) Clinical Commissioning Group (CCG)
* Age 18-49
* Not previously invited for COVID-19 vaccination

Exclusion Criteria:

* Patients who have notified their GP that they wish to decline the COVID-19 vaccination.
* Patients' whose medical records report a severe allergy to medicines (as per the JCVI guidance)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120000 (Estimated)
Dates: Start 2021-05-11 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-11 (Estimated)

PRIMARY OUTCOMES:
COVID-19 vaccination uptake at 3 weeks | 3 weeks from invitation text message
  COVID-19 vaccination uptake at 3 weeks

SECONDARY OUTCOMES:
COVID-19 vaccination uptake at 8 weeks | 8 weeks from invitation text message
  COVID-19 vaccination uptake at 8 weeks
COVID-19 vaccination uptake by demographics | 3 and 8 weeks
  Exploratory analysis of COVID-19 vaccination uptake by demographics (age, gender, IMD decile, ethnicity, previous flu vaccination)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Huf, MBBS PhD, Principal Investigator — Imperial College Health Care Trust

IPD SHARING:
Plan to Share IPD: No
The data is only available through the WSIC dataset through a de-identified dataset platform. The get access to this platform, researchers would need to get approval through the usual process to be able to access the data. The de-identified dataset cannot be exported from this trusted research environment.

REFERENCES:
- [Derived] Huf SW, Grailey K, Crespo RF, Woldmann L, Chisambi M, Skirrow H, Black K, Hassanpourfard B, Nguyen J, Klaber B, Darzi A. Testing the impact of differing behavioural science informed text message content in COVID-19 vaccination invitations on vaccine uptake: A randomised clinical trial. Vaccine. 2024 Apr 19;42(11):2919-2926. doi: 10.1016/j.vaccine.2024.03.059. Epub 2024 Mar 28. PMID 38553291